## **STUDY TITLE:**

# Effect of Tao calligraphy Meditation and Energized Water on Depression

Randomized Control Cross-over Study

### PRINCIPAL RESEARCH INVESTIGATOR:

Name: Peter Hudoba, MD, FRCS

Department: Sha Research Foundation, San Francisco, California

## PRINCIPAL CLINICAL INVESTIGATOR:

Name: Laurie Omuro-Yamamoto, PsyD, PhD Satori Family Wellness Center, Maui, HI laurieoy@gmail.com

## **VERSION DATE:**

Version 1 of 20th February 2021

### **RELATED STUDIES:**

None

## 1.0 Purpose and rationale of the study:

#### **OBJECTIVES**

The study is intended to measure the effects and determine the efficacy of Tao Calligraphy mindfulness practice on Depression. In our previous studies, the participants that regularly practice have reported a decrease in symptoms of their illness as perceived subjectively, an improvement in laboratory results or other tests and observed signs of progress reported by treating clinician and expressed an increase in well-being as measured by standardized scientific questionnaires.

#### **HYPOTHESIS**

The research hypotheses are that individuals with unipolar depression who receive energy transmission (blessing) for their affliction, who will regularly practice meditations with Tao Calligraphy and drink energized water will report:

- 1) a decrease in the symptoms of their illness as perceived subjectively.
- 2) an improvement of the clinical status of their illness, as observed by their clinicians.
- 3) improvement of well-being or clinical status as measured by standardized scientific questionnaire (s).

#### **BACKGROUND**

Chinese calligraphy handwriting is a dynamic process of integrating visual spatial awareness, cognitive planning and motor skills that is maneuvered with a brush to follow defined configurations of characters. [1]. There has been growing empirical studies of Chinese calligraphic handwriting that resulted in improvements in visual attention and span, increased mental concentration [2], confirming it as an effective treatment for psychosomatic conditions and post-traumatic hyperarousal symptoms [3] and exhibited significant effects on hypertension and type 2 diabetes [4] [5]. Leisure activities occurring later in life that includes calligraphy may inhibit cognitive decline [6].

Tao Calligraphy is a unique branch of Chinese calligraphy (Yi Bi Zi) in that it is characteristic of one stroke writing. Every character is written with one continuous stroke with the brush always in contact with the paper. [7] Results from studies confirmed efficacy in tracing in post-acute rehabilitation setting in that patients reported being less incontinence, shortened duration of hospital stay, an increase in overall well-being. [8] Retrospective analysis of data exhibited improvement in general wellbeing, an increase in optimism and energy level, as well as improvement of their symptoms. [9] According to a study measuring the effects of calligraphy tracing meditation with mantra chanting (repeated sound or word to aid with concentration saying out loud or silently) of spiritual practitioners, the results exhibited statistically positive improvement in Physical Functioning, Role Limitations due to physical health problems; Role Limitations due to Personal or Emotional Problems; Energy / Fatigue; Emotional Well-

being; Social Functioning; Bodily Pain; General Health. [10] In the prospective follow up study of these subjects, following 6 months they continued to improve in functioning in the above-mentioned areas. The authors concluded that tracing calligraphy and mantra chanting was simple to follow, well tolerated and no complications arose during the study. [11]

Medical conditions, life threatening diseases, degenerative illness and mental health challenges impairs functioning that interfere with activities of daily life, and negatively impacts overall well-being. Current studies suggest that life expectancy of an individual decreases with each additional chronic condition. [12] Individuals diagnosed with major depressive disorder are susceptible for cardiovascular disease and stroke. [13] Following a heart attack, people experiencing depression increases their risk for cardiac-related death three-fold. Also, diabetes doubles the risk for depression. [14] Well-being incorporates mental health (mind) and physical health (body) that results in more holistic interventions for disease prevention and health promotion. [15] Cross-sectional, longitudinal and experimental studies indicate that well-being is associated with Self-perceived health, Longevity, Healthy behaviors, Mental and physical illness, Social inter-connectedness, Productivity and Factors in the physical and social environment. [16] [17]

#### 2.0 RATIONALE

The study aims to acquire both basic and applied knowledge to which the primary purpose is gain the measurable data of individuals with various illnesses to meditation with Tao Calligraphy, specifically focused on the alleviation of their condition. Thus, proposing another method of rehabilitation that would be integrated into their conventional medical treatment and care.

#### THEORETICAL FRAMEWORK

Tao Calligraphy art has been studied in the US and Canada since 2013, producing significant results in improving overall well-being and an efficacious intervention for individuals with chronic conditions. This is a unique style of moving meditation, where mindfulness (heightened awareness) is achieved by the combination of movement and focus on Calligraphy art. In this practice, the subjects trace the lines of calligraphy with fingers and simultaneously say loudly or silently an affirmation (mantra), which enables them to achieve deep concentration during wakefulness. The proposed research to measure the effects of Tao Calligraphy will further provide collective data to offer an integrative intervention for individuals seeking additional treatment that is of minimal risk and to maximize benefits to address condition.

The proposed research is focused on the effects of transmission of pure energy (blessing) and meditation on humans with a specific illness or health condition.

This study is a fully developed project, based on experiential data obtained from several previous pilot and formal studies.

The soul healing techniques of the Power Healing system were evaluated in a "Cancer Recovery Pilot Study" conducted from November 1, 2000 to February 14, 2001. This study was led by Master Sha and John Gray, and Elizabeth Targ MD as a director. It was approved by the internal board of the Complementary Medical Research Institute (CMRI) and the California Pacific Medical Center (CPMC), San Francisco. This study employed Western psychological techniques with Eastern energy balancing techniques. An analysis of the data from the Pilot Study confirmed the validity and efficacy of Zhi Neng Medicine and Power Healing techniques in the treatment of cancer. A statistically significant improvement of Karnofsky and EORTC scores was observed upon completion of the three-month program.

The effect of Zhi Gang Sha's transmission of a pure energy (blessing) was also evaluated in the "Change of the Heart Double Blind Randomized Crossover Study" conducted from August 15 to October 10, 2005.

This study was approved by the internal board of Sha Research Foundation in San Francisco The initial results of the study confirmed that it is possible to measure the effects of a long-distance blessing on the energy and spiritual systems of recipients. Some of the changes measured were statistically significant. Analysis of data from the study showed statistically significant improvements in empathy, egotism, mental and emotional well-being, and the quality of meditative states. Some (but not all) remote viewers were able to document changes in the spiritual images, producing statistically significant differences between blessed and control groups. Regression analysis showed dependency on the length and depth of the spiritual practice of subjects.

The effects of Zhi Gang Sha's transmission of pure energy (blessing) and meditations were also evaluated in the "Miracle Healing Case Studies," conducted from November 2013 to November 2016 (Level 1) and from 2017 until 2021 (Level2) and from 2019 until now (Level 3).

These studies were approved by IRB at Aurora, ON, Canada. The Level 1 study was completed successfully and most of the subjects who did participate in the study until its conclusion reported marked reduction of symptoms and no side effects from the practices. The results were presented at several conferences in the USA. In Level 2 study, the subjects reported marked reduction of symptoms and no side effects from the practices. Statistical analysis of the research questionnaire was significantly positive. The results were presented at several conferences in the USA. The subjects in Level 3 study also reported marked reduction of symptoms and no side effects from the practices. Statistical analysis of the research questionnaire was significantly positive. The results were submitted for presentation at upcoming conference in the USA.

No risks or negative side effects of the transmission of pure energy given to human participants or meditation with Tao Calligraphy have been observed in these pilot projects and formal studies.

For the list of Research Presentations please refer to Appendix A.

#### **METHOD**

This study will determine the effects of transmission of a pure energy (blessing), meditation with Tao Calligraphy and drinking energized water as measured through subjective and objective evaluations of changes in depression in the subjects.

## **Design of the Study**

The study will be performed as a Randomized Controlled Cross-over Trial. New subjects may enter the study at any time. After new subjects are admitted into the study, they will be randomized into either the treatment or the control group.

All subjects that are randomized into the **control** group will be observed only (without doing any practice) during the 1<sup>st</sup> six weeks. They will then be switched into the treatment group, will receive a transmission of a pure energy (blessing) and will be practicing Tao meditation, and drinking energized water daily for the 2<sup>nd</sup> six weeks.

All subjects that are randomized into the **treatment** group will receive a transmission (blessing) and will be practicing Tao meditation and drinking energized water daily during the  $1^{st}$  six weeks. They will then be switched into the control group and will be asked to stop any meditation for the  $2^{nd}$  six weeks.

Every subject who is accepted into the study, will receive transmission (blessing) by Zhi Gang Sha (or his designee) prior to the commencing meditation practice, will be instructed on how to practice meditations with Tao Calligraphy and how to energize the water they will drink.

New subjects may enter the study at any time. After new subjects are admitted into the study, they will be randomized into either the treatment or the control group and analyzed at monthly regular intervals for two months.

#### **Data collection:**

Participants in both control and treatment group will complete the questionnaire (s) at the entry time point (Time 0), at the end of  $1^{st}$  six weeks (Time 1), and at the end of  $2^{nd}$  six weeks (Time 2).

Every subject who is accepted into the study, will receive prior to the inception of practice transmission of pure energy (blessing) and will be instructed on how to practice meditations with Tao Calligraphy, how to energize the water during this practice and to drink it.

This study will evaluate the effects of the transmission of pure energy (blessing), meditation with Tao Calligraphy and drinking energized water as follows: The study is conducted on an outpatient basis and includes:

- a telephone discussion (clarification of inclusion / exclusion criteria)
- signing of the consent /Information; instruction in the study design and practicing the Tao Calligraphy-tracing meditation and energized water drinking; first data collection questionnaires (Time 0)
- regular weekly meditation practices on Zoom with participants in the treatment
- Completion of the questionnaires by the participants at Time 1 (6 weeks) and Time 2 (at 12 weeks)
- Completion of assessments by a Study principal co-investigator

## B) Improvement of general well-being or clinical well-being as measured by standardized questionnaires (in 6 weeks intervals).

These questionnaires will be used in the study:

- 1. John Ware's SF-36 Quality of Life questionnaire
- 2. PHQ9 Depressive Symptoms (Psychometric questionnaire)
- 3. BAI-21 Beckman Inventory (Psychometric questionnaire)

All participants will complete the first questionnaire Quality of Life (SF36), PHQ9 Depressive Symptoms and BAI-21 Beckman Inventory upon entry into the study (Time 0) and then again after first 6 weeks (Time 1) and again after second 6 weeks (Time 2 - the end of participation in the study).

Transmission of pure energy and instruction of subjects on how to practice meditations with Tao Calligraphy and drinking energized water will be the sole responsibility of Universal Soul Service Corp.

Collection, handling, and evaluation of medical records and questionnaires and presentation of the research results will be the sole responsibility of Sha Research Foundation.

#### **Study Execution**

The study will be performed by collecting enrollment data and medical data directly from patients personally, over the phone, via email or on-line (Zoom). The research Questionnaires will be filled on-line using personal ID Codes – to ensure confidentiality. The codes will be emailed by the PI to each of the participants individually.

The transmission of the blessing will be conducted by Tao Academy team, who will offer the blessing to subjects of the study remotely.

Tao Academy team will be responsible for teaching subjects the meditation with Tao Calligraphy.

The transmission of pure energy (blessing) will be done to participants for free by Tao Academy certified teacher. There will be no fees for the teaching on how to meditate nor for any other aspect of participation in the study.

A copy of Tao Calligraphy Greatest Love by Dr. Zhi Gang Sha will be provided electronically.

Conversely, participants will receive no remuneration for participating in the study. Data collection, data handling, and data assessment will be the responsibility of the Sha Research Foundation's research team members who have a medical, nursing, and/or scientific background, and will be performed through personal delivery, by email and online collection.

Members of the research team will NOT administer any transmission of pure energy (blessing), teaching, or any form of medical support to participants of the study.

Participants of the study will be required to self-meditate using the Tao Calligraphy for thirty minutes every day and to record the length of practice and responses during and after each practice. They will also energize a 1 L of regular drinking water using this practice and will drink it over the course of the day to their leisure. Besides individual meditations on their own, participants will attend once a week 30 min long group meditation practice led by an Instructor, done over the Zoom.

Meditation with Tao Calligraphy instruction sheet and instruction how to energize the water will be provided to the participants. Participants will be responsible for obtaining their drinking water (either tap water or bottled water).

Process for energizing the water: Subjects will obtain 1 L bottle of their choice to which a one-time transmission of a pure energy will be given at the same time as they are receiving energy transmission to facilitate their meditation practice. Participants will fill the bottle daily with the drinking water (tap or purchased bottled water) before starting their meditation. At the beginning of meditation practice, the subject will ask to have the water energized by their meditation practice. After the meditation practice, they will drink the water throughout the day.

Subjects in the study should continue to follow their physicians' advice and recommendations during their participation in the study and should continue to receive any, and all conventional treatment in which they have been participating prior to entry into this study.

Sha Research Foundation will clearly inform participants that the teaching and research teams are not offering any medical diagnosis, guidance, evaluation, or treatment and that participation in the study is not a replacement for any conventional medical treatments or diagnosis.

Participants are also encouraged to continue their usual spiritual practices in which they have been participating prior to the study.

Participants of the study will be responsible for obtaining copies of their medical records from their medical practitioners and delivering them to Foundation officers.

The study will commence in 2021 and will last for about 3 years. The plan is to accept new subjects into the study at any time from its commencement in 2021 up to 3 September of 2024 – with expected conclusion in December of 2024.

There is no limit to the number of subjects that may be admitted to this study during the study years. Subjects can withdraw from the study with no penalty at any time for whatever reasons they may have.

## 3.0 Enrollment Criteria (who can be in your study and who would not be eligible to participate in your study):

### **Patient Population**

- 1. Subjects with diagnosed Unipolar Depression an Improvement of Depression symptoms when practicing Tao calligraphy tracing meditation and drinking energized water.
- 2. Improves the quality of life and well-being of unipolar depressive Subjects through regular Tao calligraphy tracing meditation and drinking energized water.

#### **Inclusion** criteria

- Adult subjects / patients (age 19 years and over) with a primary diagnosis as one Unipolar depression according to ICD-10 criteria is present and diagnosed by a licensed physician.
- Disease duration at least six months.
- Willingness and ability to comply with data collection requirements.
- Complete submission of required documentation prior to enrollment into the study, including informed consent and consent to release of information.
- Willingness to allow their data to be used for research purposes and published as deemed fit (while conforming to all applicable privacy laws) by Sha Research Foundation.
- Willingness to practice the daily calligraphy meditations and follow the protocol.

#### **Exclusion criteria**

- Not meeting any of the inclusion criteria
- Bipolar disorders, schizophrenia (psychosis)
- Treatment with highly potent neuroleptics
- inability to sign consent and follow instructions
- Acute suicidality, suicide plans or suicide attempts in the current disease episode or suicide attempt within the last 3 years
- Unwillingness to participate in data gathering
- Unable to follow the practice regimen, including the daily calligraphy meditations
- Pregnant or nursing. Participants who become pregnant during the study will be required to end their participation.
- Serious mental disorders (e.g., schizophrenia)
- There are no exclusion criteria placed upon potential subjects related to national origin,

culture, ethnicity, race, sex, physical disability, sexual orientation, religion, or spiritual practices.

## 4.0 Sample Size:

#### A/ Sample Size:

The study will be conducted as a randomized controlled trial. It will Subjects / patients who are between 19 and 63 years old at the time of the examination, with clinically relevant and unipolar depression (according to ICD-10, 2015) in two groups divided randomly.

The number of cases calculated was N = 55 (rounded up to 56) for both groups with one calculated drop-out rate of 15%, calculated. Here, the two-sample (two-sample) t-test applied.

#### 1<sup>st</sup> six weeks:

Assuming a symptom reduction of 30% in group I and 0% in group II and a standard deviation of 30%, you need 90% power 23 patients per group, for a total of N = 46.

#### 2<sup>nd</sup> six weeks:

The same number of cases results after the second month. If one goes from one Symptom reduction of 60% in group I and 30% in group II and one Standard deviation of 30%, with a power of 90% you need 23 patients per Group, that is a total of N = 46.

Taking into account a drop-out rate of 15%, in both cases N = 55 (rounded up to 56) patients needed.

Group I: Tao calligraphy mediation group I (number 28)

Group II: Control Group II (number 28)

The evaluation of Quality of Life and Psychometric questionnaires is done by means of the program PSPP using appropriate parametric and non-parametric tests: For statistical analysis of scores obtained from questionnaires we will use Anova, two-way Anova and regression analysis, we set confidence level at 95%.

The results of the study will be published on the Foundation website and on the scientific meetings and journals. The audience is expected to be the health care, scientific, and integrative, complementary, and alternative medicine communities.

The data and results of the study remain the intellectual property of Sha Research Foundation.

#### Authorship of the data of this study will be based on:

- 1. degree of contribution to the conception or design of the study
- 2. degree of creating any important intellectual content of the study
- 3. degree of participation on creating final report

4. an agreed role in the conduct of the study.

## 5.0 Recruitment and Screening Methods:

Recruitment announcement with be placed at:

Sha research foundation website: www.ShaResearchFoundation.com

Sha Research Foundation Twitter and Facebook

Social media Depression Support groups

Letters in selected psychiatric and psychologist offices

Advertisement in newspaper and magazines.

We are submitting previously approved letter and advertisement for the study Pro00031067.

#### **SCREENING METHODS:**

- **1)** Diagnosis must be made by a licensed medical professional a specialist in the field, outlined in a formal medical letter with clinical symptoms, signs, and results of tests at the time diagnosis was made.
- **2)** Medical reports as applicable to the given illness, at the time diagnosis was made.
- **3)** Research data by standardized questionnaire collected at the time of entry to study and at the times of 6-week follow up intervals.

#### 6.0 Research Locations:

Satori Family Wellness Center 339 Kalua Road, Wailuku, HI 9679 Phone: 808.205.6637

## 7.0 Multi-site Research (research that involves external collaborating institutions and individuals):

| N/A |
|-----|

## 8.0 International Research (where data collection will occur outside the United States and U.S. territories, including online activities)

The research will take place in the U.S.A and Canada only.

#### 9.0 Procedures Involved:

The study is conducted on an outpatient basis and includes:

• A personal or telephone discussion (clarification of inclusion / exclusion criteria) signing of the consent /Information;

- instruction in the study design and practicing the Tao Calligraphy-tracing meditation and energized water drinking;
- first data collection questionnaires at Time 0
- randomization into intervention and control groups
- regular Zoom practices with participants in the intervention group (or pre-recorded meditation practices with certified teachers as a back-up)
- Completion of the questionnaires by the participants at Time 1 (6 weeks)
- Cross-over after completion of 1<sup>st</sup> six weeks (intervention group becomes a control group, and control group becomes intervention group)
- Completion of the questionnaires by the participants at Time 2 (at 12 weeks)
- Completion of assessments by a Study principal co-investigator

Procedures to protect subjects who are found to be at risk of self-harm during the study:

- a. All subject will be required continue their conventional medical treatment and support with their health care providers.
- b. Subjects will be notified during initial interview that the participation in the study does not offer any diagnosis and does not replace convention treatment.
- c. We require that the participants continue to be under the medical supervision of their health care providers.
- d. Clinical PI is licenced psychologist in the USA who will be reviewing the questionnaires right after they were filled up to identify if the results do not represent a risk of suicide in the subjects
- e. At the time of screening participants will be given the phone number to the clinical investigator where they can call in the time of distress.

| 10.0 | Research with Vulnerable Populations (if children are the ONLY |
|------|----------------------------------------------------------------|
| | vulnerable population you plan to enroll, do NOT complete this |
| | section instead fill out Appendix A) |

| N/A |
|-----|

## 11.0 Incomplete Disclosure or Deception:

N/A

#### 12.0 Consent Process:

Trained research team member(s) will follow SRF Consent process V1.0 20200306. After obtaining the name and contact of potential participant from the PI, research team member will connect with the potential subjects for screening using inclusion and

exclusion criteria of the study. This will be done either in person, over the phone or Zoom meeting. If the consent is done by the phone-call or Zoom, signature will be issues on behalf of the participant by the consenting research team member and witnessed by a second person. Participant will be given a copy of the consent form and a study information letter for the participants, explaining the study in more detail. For consent form see Main ICF.

The signed consent will be sent to and stored at Sha Research Foundation for 7 years.

## 13.0 Waiver of Participant Signature on Consent Form:

We would like to apply for a waiver of documentation of consent for verbal consent so that consent can be obtained remotely.

#### 14.0 Waivers and Alterations of Consent Information:

N/A

## 15.0 Financial Compensation:

There will be no compensation of research participants.

Participants may incur cost related to copying or faxing documents.

Participants will receive free instructions and weekly practices with instructor.

Participants will receive free transmission of pure energy (blessing).

Research involves Minimal Risk to the participants; therefore, no compensation will be available to the participants.

## 16.0 Audio/Video Recording/Photography

We will not be performing any video, audio or photography recording.

#### 17.0 Potential Benefits of this Research:

There has been growing empirical studies of Chinese calligraphic handwriting that resulted in improvements in visual attention and span, increased mental concentration, confirming as an effective treatment for psychosomatic conditions and post-traumatic hyper-arousal symptoms, and exhibited significant effects on hypertension and type 2 diabetes. Leisure activities occurring later in life that includes calligraphy may inhibit cognitive decline. Our own studies clearly documented improvement in Wellbeing Scores (Rand SF-36

questionnaire), improvement in pain scores (McGill pain questionnaire) in subject suffering from chronic pain. Improvement in depression scores (BDI, PHQ9 and HAM questionnaires) in patient with depression. Wellbeing and pain study has been already presented at the conference. Depression study (from Germany) was recently submitted for presentation.

## 18.0 Potential Risks to Participants:

No risks or negative side effects of the blessings given to human participants or calligraphy meditation with Tao Calligraphy have been observed in our pilot projects and formal studies.

## 19.0 Provisions to Protect Participant Privacy and Data Confidentiality:

All scientific data will be stored in the computer in spreadsheet under ID code numbers according to Tri Council Policy Statement: Ethical Conduct for Research Involving Humans (2005).

A unique ID code number will be assigned to each participant for entry for internal tracking. Once the unique ID number is assigned, no personal identity information is kept with research spreadsheets.

The data collected via website will have only confidential ID assigned and never any names or personal identifiers. As there are no names associated with participants' responses in their electronic research files, it would be impossible to know which subject these responses belong to.

When client provides medical or personal information in paper form, these are scanned and forwarded to research team by email. Paper original documents are returned to participant who provided them. Once the email with documents is received by research team, downloaded to research external hard drive, and confirmed receipt, the emails with files are deleted from email inbox.

All collected personal and medical information is stored on external hard drive that can be accessed only through a password-protected Linux-based program.

There will be no hard copies of data printed out, although the results of statistical tests and actual papers for presentation will be in paper form.

## **20.0** Data Monitoring Plan to Ensure the Safety of Participants:

The collected data will remain the property of Sha Research Foundation and only members of the research team will have the access to the research data collected.

Each participant will complete an Application Form. The signed consent forms will be faxed to the Foundation. Data collection will be executed at 6-week intervals after receiving the energy transmission for total of 3 months.

#### Research Data

At the time of admission to the study, participants will provide following:

- 1) Copies of their medical records that must include a medical letter from their physician or specialist documenting the onset of their illness, symptoms, and signs, results of all relevant tests, medical procedures, and medications, and progress of the illness, at or soon after the transmission of blessing by Zhi Gang Sha (or his designee), and then again when new relevant information arises.
- 2) Participants will as well provide a letter with their subjective description of symptoms prior to the incept of Tao calligraphy meditation practice.
- 3) Participants will complete following research questionnaires prior to the incept of Tao calligraphy meditation practice, transmission of pure energy (blessing) and drinking energized water: Rand Quality of Life (SF36), PHQ9 Depressive Symptoms, BAI-21 Beckman Inventory.
- 4) During the time of the study, participants will provide the following:
- A) The medical letter from their physician or specialist documenting any change of their illness, symptoms, and signs, results of all relevant tests, medical procedures, and medications at any time when new relevant information arises.
- B) Follow up research questionnaire (our design Form 5), Rand Quality of Life (SF36), PHQ9 Depressive Symptoms, BAI-21 Beckman Inventory filled at six weeks (Time 1) and 12 weeks (Time 2) follow ups.

Standardized research questionnaires are collected at the time of entry to the study and at the times of six weeks follow up intervals, together for 3 months.

C) Data Processes

There will a Consent Process form filled after consenting procedure, this will be reviewed.

All applications are audited for completion.

The log of adverse events will be maintained (this would include data issues also).

The other logs would be: Protocol deviation Log, Subject withdrawal and termination log, Subject visit log spreadsheet, Telephone log.

Application, consent and any medical documents will be scanned and stored on large (not flash drive) external drive by principal investigator. After he confirms receipt, any person obtaining these documents will delete them from their computers and from email inbox. Once principal investigator downloads the data from inbox to a hard drive, any email containing data will be deleted from the inbox.

Research Data collected on password protected entry on the website, will have only first name

and confidential ID as identifiers, and so even in unlikely event of breach to website, no research data could be attributable to a particular person.

All data will be stored for 7 years and will be safely deleted afterwards. Any retiring hard drive will be not only erased, but also physically damaged so could not be read from anymore (in accordance to Canadian Medical Protective Association guidelines).

## 21.0 Long-term Data and Specimen Storage and Sharing:

All scientific data will be stored on external hard drive at least 7 years under ID code numbers according to Tri Council Policy Statement: Ethical Conduct for Research Involving Humans (2005) and HIPAA. All data will be deleted after 7 years.

No personal or attributable medical data will be shared outside of Sha Research Foundation.

## **22.0** Qualifications of Research Team to Conduct the Research:

Peter Hudoba, MD, FRCS, neurosurgeon, affiliated as researcher with, and prior CEO of Sha Research Foundation. Previously as a Professor of Neurosurgery, University of Saskatchewan. Mailing address: Mt Seymour Clinic, 2<sup>nd</sup> Floor, 333 Mt Seymour Boulevard, North Vancouver, BC

Laurie Omuro-Yamamoto PhD, Licensed Psychologist: Satori Family Wellness Center 339 Kalua Road, Wailuku, HI 9679 Phone: 808.205.6637 laurieoy@gmail.com
Marie-Louise Zurbach: retired medical laboratory technician; quality assurance auditor, Quebec, Canada

Rya Joy Baligad: Physiotherapist, Maui HI, U.S.A.

Anette Omuro: certified Tao academy teacher, Maui HI, U.S.A.

Nishat Kazi student of psychology with extensive experience in psychology research.

University of Toronto, Toronto, Canada

## Appendices and additional documents:

| Appendix A: SRF Research Conference<br>Appendix B: References<br>Appendix C: CVs<br>Informed Consent Form<br>Information Letter to Subjects | es Presentations 2001-2021 |
|---|---|
| Rand SF 36 Questionnaire | |
| PHQ9 Depressive Symptoms | |
| BAI-21 Beckman Inventory | |
| Allan Chuck President and CEO Sha Research Foundation | Date |
| Peter Hudoba Principal Research Investigator | Date |